CLINICAL TRIAL: NCT03366233
Title: The Role of Brain Activation and Cerebral Blood Flow in Mental Fatigue.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MF-MRI
Record Dates: First submitted 2017-12-01; First posted 2017-12-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Mental Fatigue; Healthy
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentally fatiguing task (Experimental): A modified Stroop task of 90 min, partitioned in 8 blocks of 252 stimuli, will be used as mentally fatiguing task.
  Interventions: Other: Mental fatigue
- Control task (Placebo Comparator): In the control task subjects will have to watch a documentary on the same computer screen as that used for the experimental trial for 90 min.
  Interventions: Other: Control

INTERVENTIONS:
Other: Mental fatigue — A modified Stroop task of 90 min, partitioned in 8 blocks of 252 stimuli, will be used as mentally fatiguing task. The Stroop task requires inhibition and sustained attention on controlled processes.
  Arms: Mentally fatiguing task
Other: Control — In the control task subjects will have to watch a documentary on the same computer screen as that used for the experimental trial. These documentaries are chosen based on their emotionally neutral, yet engaging content.
  Arms: Control task

SUMMARY:
To assess the changes in brain activation and cerebral blood flow due to mental fatigue in a placebo-controlled study. More specifically we want to assess whether brain activation [measured with Blood Oxygen Level Dependent (BOLD) functional resonance imaging (fMRI)] is decreased during a Flanker task in a mentally fatigued state and whether this coincides with a decline in cognitive performance. In addition we also want to evaluate whether cerebral blood flow [measured with arterial spin labeled (ASL) fMRI] in a resting state is reduced when mentally fatigued.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (No neurological/cardiorespiratory/psychological disorders)
* No medication
* Non-smoker
* Between 18 and 35 years old

Exclusion Criteria:

* Injuries
* Illness
* Pacemaker, neurostimulator, medication pump or metal implants
* Use of medication or any kind of drugs
* Use of alcohol, caffeine and heavy efforts 24 hours before each trial
* Not eating the same meal the night before and the morning of each trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent - Signal during a 10-min cognitive task (i.e. Flanker task) | Blood Oxygen Level Dependent - Signal will be measured during a 10-min Flanker task that will be completed immediately prior and after the 90-min task that is completed in both trials.
  Blood Oxygen Level Dependent - Signal will be measured during a 10-min Flanker task that will be completed immediately before and after the 90-min task (i.e. documentary in control trial; stroop task in intervention trial)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Physiology and Sports Physiotherapy Research Group, Brussels, (non-US), Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Cutsem J, Van Schuerbeek P, Pattyn N, Raeymaekers H, De Mey J, Meeusen R, Roelands B. A drop in cognitive performance, whodunit? Subjective mental fatigue, brain deactivation or increased parasympathetic activity? It's complicated! Cortex. 2022 Oct;155:30-45. doi: 10.1016/j.cortex.2022.06.006. Epub 2022 Jun 30. PMID 35964356